CLINICAL TRIAL: NCT07038499
Title: Prevalence and Determinants of Migraine Among Headache Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Foo Chai Nien, Assiociate Professor, Universiti Tunku Abdul Rahman
Other Study IDs: 2024[K]122; 2024[k]-122 (Other: Hebei University of Engineering Affiliated Hospital)
Record Dates: First submitted 2025-05-23; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Headache (Migraine)
Keywords: Pain; Headache; Migraine; Disability
MeSH Terms: conditions — Migraine Disorders; Pain; Headache

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:  — Participants are not assigned an intervention as part of the study.

SUMMARY:
Migraine is a prevalent and disabling neurological condition that often coexists with other health issues, such as hypertension and impaired physical, mental, and social functioning. Understanding the prevalence of migraine and its associations with these health domains can provide valuable insights into the broader impact of migraine on overall well-being. By focusing on patients at the Affiliated Hospital of Hebei University of Engineering in China, this study can identify specific health burdens within this population, inform integrated clinical management strategies, and support the development of targeted interventions to improve patient outcomes and quality of life.

DETAILED DESCRIPTION:
Migraine is a common and disabling neurological disorder that poses a significant public health burden worldwide. In China, the estimated prevalence of migraine is approximately 9.3%, with higher rates reported among women and individuals of working age. Despite being one of the most prevalent types of primary headache disorders, migraine remains underdiagnosed and undertreated in many regions of China, partly due to limited awareness and access to specialized care. Concurrently, hypertension is highly prevalent in the Chinese adult population, with nearly one in four adults affected, making it a leading contributor to cardiovascular morbidity. Emerging evidence suggests a potential bidirectional relationship between migraine and hypertension, possibly linked through shared pathophysiological mechanisms such as endothelial dysfunction, autonomic dysregulation, and inflammatory pathways.

Moreover, migraine is often associated with detrimental effects on physical, mental, and social health, including impaired physical function, increased pain intensity, depression, anxiety, fatigue, sleep disturbances, and reduced ability to participate in social roles and activities. However, studies exploring these multidimensional impacts in Chinese clinical populations remain limited.

Therefore, this study aims to investigate the prevalence of migraine and its association with hypertension as well as physical, mental, and social health domains among headache patients at the Affiliated Hospital of Hebei University of Engineering, China.

ELIGIBILITY:
Inclusion Criteria:

• Patients diagnosed with headache according to the International Classification of Headache Disorders, 3rd Edition (ICHD-3).

Exclusion Criteria:

* Patients with other major diseases or severe mental disorders;
* History of endocrine, immune, or nervous system diseases or other severe somatic diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending at the Affiliated Hospital of Hebei University of Engineering, China.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Estimated)
Dates: Start 2025-06-23 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of migraine | Day 1
  The overall number and proportion of people with migraine (according to the International Classification of Headache Disorders, 3rd edition (ICHD-3))

SECONDARY OUTCOMES:
Correlation with hypertension | Day 1
  Hypertension will be assessed using self-reported hypertension status (Yes/ No)
Correlation with physical (physical function, pain intensity)， mental (depression, anxiety, fatigue, sleep disturbance) and social (ability to participate in social roles and activities) | Day 1
  Patient-Reported Outcomes Measurement Information System (PROMIS) measures domains including physical (physical function, pain intensity)， mental (depression, anxiety, fatigue, sleep disturbance) and social (ability to participate in social roles and activities). The total score of each domain is converted to a standardized T score. High scores mean more of the domains being measured.
Correlation with migraine disability | Day 1
  The MIDAS (Migraine Disability Assessment) is a validated questionnaire used to measure headache-related disability over the past three months. It consists of five questions, each addressing the number of days affected by migraines. Each answer is recorded as a number of days. The higher score indicating more severe migraine disability
Correlation with quality of life | Day 1
  The Migraine-Specific Quality of Life Questionnaire (MSQ) is a validated tool used to assess the impact of migraine on a patient's quality of life. Raw scores are first calculated by summing item responses for each domain. Raw scores are then transformed into a 0-100 scale, where higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Chai Nien Associate Professor, PhD, Principal Investigator — Universiti Tunku Abdul Rahman
Locations (1):
- Affiliated Hospital of Hebei University of Engineering, China, Hebei, China

IPD SHARING:
Plan to Share IPD: No